CLINICAL TRIAL: NCT05698940
Title: Subjective and Objective Outcome of Septoplasty With or Without Infundibulotomy/Uncinectomy
Brief Title: Subjective and Objective Outcome of Septoplasty With or Without Infundibulotomy
Acronym: InfundSPL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: KEK 2015-0356
Record Dates: First submitted 2022-12-27; First posted 2023-01-26 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Nasal Blockage; Nasal Obstruction; Septum; Deviation
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infundibulotomy (Active Comparator): Infundibulotomy on one side of sinuses
  Interventions: Procedure: Infundibultomy
- No Infundibultomty (Sham Comparator): No Intervention on other side of sinuses
  Interventions: Procedure: Infundibultomy

INTERVENTIONS:
Procedure: Infundibultomy — Infundibultomy on one side of patient

SUMMARY:
Septoplasty is one of the most common procedures in rhinology. In many centers and private institutions, an infundibulotomy is performed in addition to septoplasty without evidence of significant improvement for the patient. Often the reason given for this is the improvement of the functional outcome in terms of better nasal breathing, although there is no evidence for this. If a significantly better outcome can be shown, one would have a first evidence for the extended procedure.

ELIGIBILITY:
Inclusion Criteria:

Unilateral breathing impairment due to septal deviation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2016-03-29 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Single sided VAS Scores for breathing impairment | 3 months
  Rating of nasal breating on a 0-10 scale

SECONDARY OUTCOMES:
SNOT Score | 3 months
  Quality of Life Measure from 0-110
NOSE Score | 3 months
  Nasal symptom questionnaire
PNIF | 3 months
  Peak Nasal Inspiratory Flow measured in ml/sec

CONTACTS AND LOCATIONS:
Locations (1):
- Zurich University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No